CLINICAL TRIAL: NCT02831140
Title: The Fast Track Rehabilitation in Thoracic Surgery - A Prospective Randomized Study
Brief Title: The Fast Track Rehabilitation in Thoracic Surgery
Acronym: FTR-TS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Habib Bourguiba University Hospital (Other)
Collaborators: Community medicine department -Habib Bourguiba University Hospital (Unknown)
Responsible Party: Principal Investigator, Abdessalem Hentati, Thoracic surgeon, Habib Bourguiba University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FTRCCVTSFAX
Record Dates: First submitted 2016-05-26; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Thoracic Surgery
Keywords: Fast track; rehabilitation; post operative complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Common arm : for both groups : (Other): * In preoperative phase
  * In peroperative phase
  * In postoperative phase
  Interventions: Behavioral: commun interventions
- FTR protocol group (A) (Experimental): A. Experimental : FTR protocol group :
  Early exercises after a thoracic surgery : removing urinary probe and all catheters as well as alimenting .
  Interventions: Behavioral: Early exercises; Behavioral: Removing urinary probe and all catheters.; Behavioral: Early alimentation
- Control group (B) (No Intervention): Traditional, conventional care group with first get up and alimentation permission in 24 hours at the postoperative.

INTERVENTIONS:
Behavioral: Early exercises — In postoperative phase:
  Early exercises: within the first hour ;setting a half bed position, deep breathing and coughing . In the second hour, curbing vagal malaise and performing relaxation movements. In the third hour, walking about 20 to 30 minutes.
  Arms: FTR protocol group (A)
Behavioral: Removing urinary probe and all catheters. — In postoperative phase : Removing urinary probe and all catheters.
  Arms: FTR protocol group (A)
Behavioral: Early alimentation — In postoperative phase :Early alimentation: in the first hour to the second hour .
  Arms: FTR protocol group (A)
Behavioral: commun interventions — * In preoperative phase: stopping smoking at least 2 weeks, hospitalization and balanced alimentation one day before the surgery.
  * In peroperative phase : no use of benzodiazepines in the anesthesia , selective intubation , maintaining vital parameters as normal and using a mini invasive surgical approach ( video thoracoscopy , video assisted thoracoscopy , thoracotomy with preservation of the posterior muscles of the chest wall
    , preservation of Serratus anterior and the front part of Latissimus Dorsi ).
  * In postoperative phase : Immediate extubation ( less than 30 minutes from the surgery end) , peridural or paravertebral or intercostal block analgesia , no use of abusive antibiotic , all analgesic drugs are permitted if there are no contraindications and physiotherapy from the 6th hour.
  Arms: Common arm : for both groups :

SUMMARY:
This prospective, randomized study is designed to evaluate the effectiveness of postoperative care pathway using the Fast Track Rehabilitation protocol (FTR) in comparison with the traditional postoperative care.

In order to conduct this study, patients having a thoracic surgery will be randomly attributed to FTR protocol group or control group.

DETAILED DESCRIPTION:
Traditionally, patients who underwent thoracic surgery have been treated with a classical protocol which include; bed rest, ambulation prohibited for 24-48 hours and starvation for several postoperative days till the recovery of bowel. Some studies reported the efficacy of early rehabilitation protocols or FTR protocols in thoracic surgery to reduce postoperative complications and to minimize hospital stay. But these studies are few and retrospective. Prospective randomized trials focuses based on the "fast track regimen" or medical fast track that interest only on the medical component .

This prospective, randomized study is designed to evaluate the effectiveness of postoperative care pathway using FTR protocol in comparison with the traditional postoperative care.

In order to conduct this study, patients having a thoracic surgery will be randomly attributed to FTR protocol group or control group.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have lung surgery during the study period after their consents are included.

Exclusion Criteria:

* Patients who have bad general state are unable to move or require a wake in the resuscitation.
* The Patients with thoracic soft tissue surgery.
* patients having mediastinoscopy, surgery of the chest wall or mediastinum.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications: Atelectasis or re-expansion failure or pneumonic infection | within postoperative 30 days
  discharge criteria:
  * Chest tube removal
  * Unassisted ambulation
  * Afebrile without major complications
  * Willing discharge

SECONDARY OUTCOMES:
Pain | in 1st hour , 2nd hour , 3rd hour , 6th hour 24th hour , 48th hour at the postoperative , within postoperative 30 days
  score measured by the Visual Analog Scale.
The Length of Hospital Stay | within postoperative 30 days
Thoracic surgery postoperative Complications | within postoperative 30 days
  During the First Admission : Prolonged bubbling
Surgery postoperative Complications : pulmonary embolism or cardiac arrhythmia or pleural empyema | within postoperative 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Imed Frihka, Professor, Study Director — Cardiovascular and thoracic surgery department - Habib Bourguiba University Hospital
Locations (1):
- Cardiovascular and thoracic surgery department - Habib Bouguiba University Hospital, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muehling BM, Halter GL, Schelzig H, Meierhenrich R, Steffen P, Sunder-Plassmann L, Orend KH. Reduction of postoperative pulmonary complications after lung surgery using a fast track clinical pathway. Eur J Cardiothorac Surg. 2008 Jul;34(1):174-80. doi: 10.1016/j.ejcts.2008.04.009. Epub 2008 May 19. PMID 18490173
- [Background] Sokouti M, Aghdam BA, Golzari SE, Moghadaszadeh M. A comparative study of postoperative pulmonary complications using fast track regimen and conservative analgesic treatment: a randomized clinical trial. Tanaffos. 2011;10(3):12-9. PMID 25191370
- [Result] Padilla Alarcon J, Penalver Cuesta JC. Experience with lung resection in a fast-track surgery program. Arch Bronconeumol. 2013 Mar;49(3):89-93. doi: 10.1016/j.arbres.2012.09.011. Epub 2012 Dec 13. English, Spanish. PMID 23245565
- [Result] Das-Neves-Pereira JC, Bagan P, Coimbra-Israel AP, Grimaillof-Junior A, Cesar-Lopez G, Milanez-de-Campos JR, Riquet M, Biscegli-Jatene F. Fast-track rehabilitation for lung cancer lobectomy: a five-year experience. Eur J Cardiothorac Surg. 2009 Aug;36(2):383-91; discussion 391-2. doi: 10.1016/j.ejcts.2009.02.020. Epub 2009 Mar 26. PMID 19324571